CLINICAL TRIAL: NCT02786212
Title: The Effects of Dexmedetomidine on Microcirculation and Other Organ Damages After Cardiac Surgeries
Brief Title: The Effects of Dexmedetomidine on Microcirculation and Surgical Outcomes After Cardiac Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201512224MINB
Record Dates: First submitted 2016-05-18; First posted 2016-05-30 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Surgical Procedure
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): Patients receiving intraoperative dexmedetomidine infusion. Infusion duration: from 10 minutes after anesthetic induction to the end of surgery.
  Interventions: Drug: Dexmedetomidine
- control (Placebo Comparator): control group, receiving same volume of normal saline infusion.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: dexmedetomidine
Drug: Normal Saline
  Arms: control

SUMMARY:
Cardiac surgery with cardiopulmonary bypass (CPB) provokes a systemic inflammatory response that can often lead to dysfunction of major organs. Activation of the contact system, endotoxemia, surgical trauma, and ischemic reperfusion injury are all possible triggers of inflammation. Previous studies demonstrated that pro-inflammatory cytokines play an important role during this process. However, very little is known about the susceptibility of the splanchnic organs to ischemic reperfusion injury. Although the incidence of intestinal complications reported to be low, the in-hospital mortality in these patients was high at 15% to 63%.

Dexmedetomidine, a highly selective α2-adrenergic agonist, can reduce the consumption of other sedative and antinociceptive drugs and provide sufficient sedative effects with minimal respiratory side effects. In addition, dexmedetomidine gradually has gained popularity in the field of critical care. Preemptive administration of dexmedetomidine has shown to be protective against inflammation, intestinal, renal, and myocardial injuries in animal and human studies. Dexmedetomidine is also used as an anesthetic adjuvant during surgery to offer good perioperative hemodynamic stability and an intraoperative anesthetic-sparing effect. Perioperative use of dexmedetomidine can reduce intestinal and hepatic injury after hepatectomy with inflow occlusion under general anesthesia. However, whether or not it can exert protective effects on the above-mentioned organs, especially intestine, after cardiac surgery remains unclear. The aim of this study is to evaluate the effects of dexmedetomidine on intestinal, hepatic, and other organ injury in patients receiving cardiac surgery with CPB.

In this double-blinded randomized controlled study, serum diamine oxidase activity, which is a sensitive and specific marker for the detection of intestinal injury, is taken as the primary endpoint. Other parameters reflecting the functions of liver (AST/ALT), lung (lung injury score and CC-16), kidney (BUN/Cre), and heart (CK-MB/Troponin T), the biomarker of endothelial injury (endocan) will also be determined. Besides, microcirculation parameters measured with Cytocam® and near-infrared spectroscopy (NIRS) will be used to estimate the protective effect of dexmedetomidine on microcirculation. The variables will be collected perioperatively and will be followed up for 3 days after the surgery. Clinical outcome parameters will be followed up for 3 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* left ventricle ejection fraction < 40%
* acute myocardial infarction within 3 months
* angina within 48 hours before surgery
* COPD
* previous history of inflammatory bowel disease
* diarrhea within 7 days before surgery
* previous cardiac surgery
* receiving non-pharmacological cardiac supportive management
* previous pulmonary embolism
* previous deep vein thrombosis
* allergic to dexmedetomidine
* refractory bradycardia (HR < 60/min )

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Perioperative changes in perfused vessel density (PVD) | 1 hours, 24 hours, and 48 hours after surgery
  PVD measured by using sublingual vital videomicroscopy

SECONDARY OUTCOMES:
Incidence of postoperative acute kidney injury | 48 hours after surgery
  Acute kidney injury diagnosed based on the KDIGO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yuan Shih, MD, Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan